CLINICAL TRIAL: NCT06437418
Title: Association of Biliary Tract Disorders in Chronic Kidney Disease Patients and Its Related Risk Factors
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, rehab Mohamed Mohamed, resident doctor, Assiut University
Other Study IDs: Gallbladder dysfunction in CKD
Record Dates: First submitted 2024-05-26; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: CKD; Gall Bladder Dysfunction
Keywords: CKD; gall bladder dysfunction; gall bladder ejection fraction; hemodialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group I: Gallbladder dysfunction in pre-dialysis CKD patients.
  Interventions: Diagnostic Test: abdominal ultrasonography.
- Group II: Gallbladder dysfunction in end stage CKD patients on dialysis.
  Interventions: Diagnostic Test: abdominal ultrasonography.
- Control Group: Gallbladder dysfunction in normal renal function participants (control group).
  Interventions: Diagnostic Test: abdominal ultrasonography.

INTERVENTIONS:
Diagnostic Test: abdominal ultrasonography. — Evaluate the gallbladder ejection fraction (EF)

SUMMARY:
Our aim in this cross-sectional study is to determine the frequency and aspects of gallbladder dysfunction and the related risk factors in pre-ESRD and hemodialysis patients.

DETAILED DESCRIPTION:
Biliary tract disorders including cholelithiasis, cholecystitis, and other diseases of the biliary tract, are one of the most prevalent medical issues in the digestive system, posing a myriad of challenges for health workers and patients. Gallbladder dysfunction is the most frequent cause of symptomatic and complicated biliary tract disorders. Although gallbladder dysfunction is a common condition in Middle East countries, data on the incidence of end-stage renal disease (ESRD) are limited. The occurrence of gallbladder dysfunction in patients fed with low-protein diets suggests that gallbladder stones formation is affected by dietary protein content. Also the lithogenic composition changes of bile, increased nucleation tendency, and impaired motility of gallbladder are important factors in ESRD patients. It has been reported that chronic kidney disease (CKD) patients on regular hemodialysis (HD) have increased bile cholesterol levels and an increased bile saturation index. In addition, the gallbladder is innervated by the autonomic nervous system, which malfunctions in uremia, and it has been shown that gallbladder stasis might cause increased stone formation. In some studies, the prevalence of gallbladder dysfunction has been shown to increase in patients undergoing hemodialysis (HD) treatment for ESRD. So, we focused in this study to try to find association of gallbladder dysfunction in pre-dialysis ESRD and HD patient in comparison to normal renal function individuals.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed as CKD with eGFR according to Cockcroft-Gault Equation, whatever they are on regular hemodialysis or pre-dialysis without history of previous gallbladder dysfunction with normal renal function individuals.

Exclusion Criteria:

* Patients who are younger than 18 years.
* Patients who are diabetic.
* Patients who have body mass index (BMI) more than 30.
* Patients who have family history of gallbladder disorder.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: individuals visiting outpatient clinics of nephrology, GIT and internal medicine in Assiut hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Gallbladder dysfunction in CKD patients | measuring fasting gallbladder volume (FV) after 10 overnight hours fasting and the residual gallbladder volume (RV) after 30 minutes after standard fixed meal
  Evaluate the gallbladder ejection fraction (EF) which will be calculated by following formula. (EF = (fasting gallbladder volume (FV) - residual gallbladder volume (RV)) / fasting gallbladder volume (FV)x 100) EF = (FV - RV) / FV x 100

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of medicine Assiut university, Asyut, Egypt